CLINICAL TRIAL: NCT02869256
Title: Regional Central Database Recording of Chronic Myeloid Leukemia
Acronym: LMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2014-LMC
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; practices evaluation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Practices evaluation — Practices evaluation

SUMMARY:
It will be a centralized database , multicentre (6 centers) , regional, chronic myelogenous leukemia cases of registration (CML) prospectively and retrospectively.

DETAILED DESCRIPTION:
Given the complexity and evolution of recommendations and to harmonize these, it appears necessary to establish a central database for recording , monitoring patients with CML supported by the participating centers the region and evaluation of care practices in use .

Indeed , the main purpose of this database is to provide diagnostic and therapeutic management of reported cases of chronic myeloid leukemia and to study the prognostic factors . The main objective is to improve significantly the percentage of patients treated adequately load in the region, in the initial stages of the disease and during its evolution.

ELIGIBILITY:
Inclusion Criteria:

* chronic myeloid leukemia Diagnosis (CML) in chronic phase , accelerated or blast
* male or female patient aged 18 years or more
* Cases transmitted by referring hematologist , one of the 6 participating centers after patient's oral information
* Clinical record presented Concertation Meeting LMC Multidisciplinary coordinated by the Institute Bergonié

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic myeloid leukemia diagnosis in chronic phase
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
compliance of the management of patients with chronic myeloid leukemia compared to the guidelines | 10 years

SECONDARY OUTCOMES:
overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Universitaire de Dax, Dax
  - Centre hospitalier Libourne, Libourne
  - Centre Hospitalier Universitaire de Pau, Pau

IPD SHARING:
Plan to Share IPD: No